CLINICAL TRIAL: NCT05634278
Title: Pilot RCT of Mindfulness Intervention in Orthopedic Trauma Patients
Brief Title: Mindfulness Intervention in Orthopedic Trauma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Adam Hanley, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB_00085446 AM_00046459
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mind wandering (Placebo Comparator)
  Interventions: Behavioral: Mind wandering
- Preoperative Mindfulness (Active Comparator): Participants will only listen to the guided meditation practice before surgery.
  Interventions: Behavioral: Preoperative mindfulness; Behavioral: Mind wandering
- Preoperative and Postoperative Mindfulness (Active Comparator): Participant will listen to the guided meditation practice before surgery and during their hospital stay after surgery.
  Interventions: Behavioral: Preoperative mindfulness; Behavioral: Postoperative mindfulness

INTERVENTIONS:
Behavioral: Preoperative mindfulness — A seven-minute, audio-guided, mindfulness meditation practice.
  Arms: Preoperative Mindfulness; Preoperative and Postoperative Mindfulness
Behavioral: Postoperative mindfulness — A seven-minute, audio-guided, mindfulness meditation practice.
  Arms: Preoperative and Postoperative Mindfulness
Behavioral: Mind wandering — A timed, seven-minute mind wandering period during which participants are instructed: "For the next 7 minutes, allow your mind to wander."
  Arms: Mind wandering; Preoperative Mindfulness

SUMMARY:
This project a single-site 3-arm parallel group randomized clinical trial conducted at a tertiary level 1 trauma center among patients undergoing operative fixation of a lower extremity fracture.

ELIGIBILITY:
Inclusion Criteria:

* Age at presentation between 18 and 65 years
* Acute lower extremity fracture to be operatively managed
* Glasgow Coma Scale of 15
* English speaking
* Willingness to participate in study

Exclusion Criteria:

* Cognitive impairment
* Pregnant or lactating woman
* Current incarceration
* Planned secondary procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Change in Preoperative Anxiety | Immediately before to after the 7-minute preoperative intervention
  Single item assessing pain unpleasantness ("How nervous, anxious, or on edge do you feel?") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater anxiety.
Change in Postoperative, In-patient Pain Unpleasantness | Immediately before to after the 7-minute postoperative intervention
  Single item assessing pain unpleasantness ("How unpleasant is your pain?") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater pain unpleasantness.

SECONDARY OUTCOMES:
Change in Preoperative Pain Intensity | Immediately before to after the 7-minute preoperative intervention
  Single item assessing pain intensity ("How much pain do you have?") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater pain intensity.
Change in Postoperative, In-patient Pain Intensity | Immediately before to after the 7-minute postoperative intervention
  Single item assessing pain intensity ("How much pain do you have?") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater pain intensity.
Change in Preoperative Pain Unpleasantness | Immediately before to after the 7-minute preoperative intervention
  Single item assessing pain unpleasantness ("How unpleasant is your pain?") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater pain unpleasantness.
Change in Postoperative, In-patient Anxiety | Immediately before to after the 7-minute postoperative intervention
  Single item assessing pain unpleasantness ("How nervous, anxious, or on edge do you feel?") scored on an 11-point (0=Not at all, 10=Very much) numeric rating scale. Higher scores indicate greater anxiety.

OTHER OUTCOMES:
Postoperative Patient Reported Outcomes Measurement Information System (PROMIS) Physical Functioning Item Bank, v2.0 | Assessed at 2-weeks, 6-weeks, 3-months, 6-months and 12-months postoperatively
  The PROMIS physical functioning computer assisted test draws from a bank of 123 items all scored on a 5 point Likert scale. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. Higher scores reflect better physical functioning.
Postoperative Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference Bank v1.1 | Assessed at 2-weeks, 6-weeks, 3-months, 6-months and 12-months postoperatively
  The PROMIS pain interference computer assisted test draws from a bank of 40 items all scored on a 5 point Likert scale. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. Higher scores reflect greater pain interference.
Postoperative Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety Bank v1.0 | Assessed at 2-weeks, 6-weeks, 3-months, 6-months and 12-months postoperatively
  The PROMIS anxiety computer assisted test draws from a bank of 29 items all scored on a 5 point Likert scale. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. Higher scores reflect greater anxiety.
Postoperative Patient Reported Outcomes Measurement Information System (PROMIS) Depression Bank v1.0 | Assessed at 2-weeks, 6-weeks, 3-months, 6-months and 12-months postoperatively
  The PROMIS depression computer assisted test draws from a bank of 28 items all scored on a 5 point Likert scale. T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points. Higher scores reflect greater depression.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States